CLINICAL TRIAL: NCT06517654
Title: Comparison of the Effectiveness of EMG-Biofeedback and Rebound Therapy in Patients With Endometriosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Çağla ÖZGÖREN, Lecturer Çağla ÖZGÖREN, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedipolU-FTR-ÇÖ-01
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Endometriosis
Keywords: Endometriosis; Pain; Quality of Life; Sleep Quality
MeSH Terms: conditions — Endometriosis; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Three parallel treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: EMG-Biofeedback (Active Comparator): In this group, pelvic floor strengthening training will be conducted with EMG-Biofeedback 2 days a week, and patients will follow a home exercise program 5 days a week. The Neurotrac® Simplex device will be used for EMG-Biofeedback. The EMG reference electrode will be placed on the patient's spina iliaca anterior superor, while two adhesive electrodes will be placed on the perineal muscles. Patients will contract and relax their pelvic floor muscles at 5-second intervals, guided by visual and auditory stimuli on the device or computer screen. Sessions will last 25 minutes, twice a week, for 8 weeks in a clinical environment. Treatment will include visual imagery for better engagement. Scores (%), and the lowest and highest EMG values (mV) will be recorded. Home exercises will be demonstrated by a physiotherapist, to be practiced 5 days a week. Patients will be instructed to report any pain during exercises to the physiotherapist.
  Interventions: Device: EMG-Biofeedback; Other: Home Exercise Program
- Group 2: Rebound Therapy (Active Comparator): In this group, rebound therapy will be performed on a trampoline, along with pelvic floor strengthening training, twice a week. Patients will also follow the home exercise program given to the first group, practicing it 5 days a week. For rebound therapy, a trampoline-based exercise program targeting pelvic floor muscles will be conducted in a clinical setting for 8 weeks, 2 days a week, with 20-minute sessions. Proper breathing patterns will be taught before starting. During rest periods, O2 saturation and maximum heart rate will be monitored. Maximum heart rate will be calculated (HRmax = 208 - 0.7 × age), and exercises will pause if it exceeds 80%. Patients will contract pelvic floor muscles during exercises, with posture corrections provided as needed. Exercise intensity will be progressively increased for adaptation. Home exercises will be demonstrated by a physiotherapist, to be practiced 5 days a week. Patients must report any pain during exercises to the physiotherapist.
  Interventions: Other: Rebound Therapy; Other: Home Exercise Program
- Group 3: Home Exercise Group (Active Comparator): Home exercise program will be taught to patients in a practical way with the physiotherapist and patients will be asked to practice at home 5 days a week. If the patient feels any pain during the exercises, they will be informed that they must report the situation to the physiotherapist.
  Interventions: Other: Home Exercise Program

INTERVENTIONS:
Device: EMG-Biofeedback — The Neurotrac® Simplex device will be used for EMG-Biofeedback treatment. As in the muscle strength assessment procedure, the EMG reference electrode will be placed on the patient's forearm, and 2 adhesive electrodes in the EMG channel will be placed on the patient's perineal muscles. The patient will be asked to contract and relax the pelvic floor muscles at certain intervals in accordance with the visual and auditory stimuli made on the device screen or computer screen. The pelvic floor muscle contraction and rest period will last 5 seconds each. The program will continue for 2 days a week, 25 minutes per session and 8 weeks and will be performed in a clinical environment. During the treatment, the treatment will be visualized for the patient with different imagery. At the end of the games played, the patients'; scores (%), the lowest and highest EMG values will be recorded in mV. The treatment will be applied to the patients in two sessions per week.
  Arms: Group 1: EMG-Biofeedback
Other: Rebound Therapy — The program will be performed in a clinical environment for 8 weeks, 2 days a week, each session will be 30 minutes. The correct breathing pattern will be taught to the patient before starting the exercises. O2 saturation and maximum heart rate will be checked during the rest periods during the exercises. The maximum heart rate will be calculated with the formula (HRmax = 208 - 0.7 × age), and the exercise will be paused when it exceeds 80%. The patient will be asked to contract the pelvic floor muscles during the exercise. Necessary warnings regarding the preservation of posture will be made throughout the exercises. The exercise intensity will be increased progressively in order to ensure the patient's adaptation to the exercises.
  Arms: Group 2: Rebound Therapy
Other: Home Exercise Program — Home Exercise Program In addition to EMG-Biofeedback Therapy in Group 1, in addition to Rebound Therapy in Group 2, and in Group 3, only a home exercise program will be applied to patients 5 days a week. The exercise program consists of diaphragmatic breathing, piriformis stretching exercise, adductor stretching exercise, gluteal stretching exercise, cat-camel exercise, happy baby position, deep squat exercise, trunk rotator stretching exercises. Each exercise will be repeated 5 times on the right and left, and 20 seconds will be waited for each repetition.

SUMMARY:
The aim of our study is to investigate the effects of pelvic floor muscle strengthening exercises with EMG-Biofeedback and pelvic floor muscle strengthening exercises with Rebound therapy on pelvic floor muscle strength, pain level, NGF level, perceived stress level, quality of life and sleep in women diagnosed with endometriosis.

DETAILED DESCRIPTION:
Endometriosis is a chronic, systematic, inflammatory, estrogen-dependent public health problem characterized by the growth of endometrial-like tissue outside the uterine cavity, including the pelvic peritoneum, rectovaginal septum and ovaries, and is particularly seen in women of reproductive age and significantly affects quality of life. The aim of our study is to investigate the effects of pelvic floor muscle strengthening exercises with EMG-Biofeedback and pelvic floor muscle strengthening exercises with Rebound therapy on pelvic floor muscle strength, pain level, NGF level, perceived stress level, quality of life and sleep in women diagnosed with endometriosis. The study will consist of 3 groups. Group 1: EMG-Biofeedback group, Group 2: Rebound Therapy Group and Group 3: Home Exercises Group. Participants will be included in the study for 8 weeks. During the evaluation, pelvic floor muscle strength will be assessed with EMG, pain level with Visual Analog Scale (VAS), perceived stress level with Perceived Stress Scale, quality of life with Endometriosis Health Profile Questionnaire (EHP-30), and sleep quality with Pittsburgh Sleep Quality Index (PSQI). NGF analysis will be evaluated by analyzing serum samples of patients with ELISA kit. Evaluations will be made before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-50 years old,
* Being diagnosed with endometriosis,
* Completing the voluntary consent form,
* Pain level being at least 4 on the Visual Analog Scale (VAS).

Exclusion Criteria:

Exclusion Criteria for the EMG-Biofeedback Group:

* Being included in another study during the study period,
* Being receiving medical treatment for endometriosis,
* Presence of gynecological bleeding,
* Presence of communication and cooperation problems,
* Presence of tubo-ovarian abscess,
* Active vaginal or urinary tract infection,
* Pregnancy and giving birth within the last 12 months,
* Presence of impaired somatosensory status,
* Not attending 2 consecutive sessions.

Exclusion Criteria for the Rebound Therapy Group:

In addition to the exclusion criteria determined for the EMG-Biofeedback Group;

* Presence of a neurological or orthopedic disease affecting the lower extremity,
* History of spine and/or lower extremity orthopedic surgery,
* Presence of severe arthritis affecting the spine and/or lower extremity,
* Presence of uncontrolled hypertension and cardiovascular disease.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women diagnosed with endometriosis are eligible to participate in the study.
Enrollment: 42 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor muscle strength | 2 weeks
  The NeuroTrac® Simplex device will be used for pelvic floor muscle strength assessment by measuring muscle activation in millivolts (mV). The assessment, performed with the patient in the lithotomy position, involves placing the EMG reference electrode on the spina iliaca anterior superior and 2 adhesive electrodes on the perineal muscles. Patients will contract and relax their muscles following auditory and visual stimuli on the screen (10 sec contraction/10 sec rest). The average, minimum, and maximum mV values will be used in the study. To ensure accuracy, measurements will be repeated 3 times and averaged.
Pain Level | 2 weeks
  Pain level will be assessed with the Visual Analog Scale (VAS), a 10 cm line from 'no pain' to 'unbearable pain,' where participants mark their pain level. The value is recorded in cm. 0 point indicates 'no pain', 10 cm indicates 'unbearable pain'.

SECONDARY OUTCOMES:
Nerve Growth Factor (NGF) Analysis | 2 weeks
  NGF levels will be analyzed using plasma samples from 3 ml blood samples. Within 30 minutes of collection, the blood will be centrifuged at 1000 x g for 15 minutes at 2-8°C. The plasma will be numbered, transferred to centrifuge tubes, and stored at -80°C until analysis. The analysis will use the Cusabio-Human NGF ELISA Kit (Catalog number: CSB-E04683h) following the kit protocol, with NGF values measured in pg/ml using a Biotek Synergy HTX device. The analysis will be repeated 3 times, and the average value will be taken. NGF sensitivity was 15 pg/ml. The Cusabio-Human NGF ELISA Kit's sensitivity range of 6.86 pg/ml-5000 pg/ml is suitable for patients with endometriosis.

OTHER OUTCOMES:
Quality of life level | 2 weeks
  Participants' quality of life will be assessed using the Endometriosis Health Profile Questionnaire (EHP-30), which evaluates health-related quality of life over the past four weeks. Scores range from 0 (best health) to 100 points (worst health).
Sleep quality level | 2 weeks
  Sleep quality will be measured with the Pittsburgh Sleep Quality Index (PSQI), covering a one-month period. Scores range from 0 to 21 points, with higher scores indicating poorer sleep quality.
Perceived stress level | 2 weeks
  Stress level will be assessed with the Perceived Stress Scale, consisting of 14 questions scored between 0-56 points. Higher scores indicate higher stress levels. Scores between 0-35 points indicate adequate stress coping, while scores between 36-56 points indicate inadequate stress coping.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Women and Children's Diseases Training and Research Hospital, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Safety Concerns